CLINICAL TRIAL: NCT06190093
Title: Safety and Effectiveness of ONS-5010 Compared to Lucentis® in Subjects with Neovascular Age-related Macular Degeneration; NORSE EIGHT
Brief Title: A 3-month Study to Assess the Safety and Effectiveness of ONS-5010 in Subjects with Neovascular Age-related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Outlook Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ONS-5010-008
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Neovascular Age-related Macular Degeneration; Age-Related Macular Degeneration; Wet Macular Degeneration
MeSH Terms: conditions — Macular Degeneration; Wet Macular Degeneration | interventions — Bevacizumab; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ONS-5010 bevacizumab (Experimental)
  Interventions: Biological: bevacizumab
- ranibizumab (Active Comparator)
  Interventions: Biological: ranibizumab

INTERVENTIONS:
Biological: bevacizumab — 1.25 mg, intravitreal injection
  Other Names: ONS-5010
  Arms: ONS-5010 bevacizumab
Biological: ranibizumab — 0.5mg, intravitreal injection
  Arms: ranibizumab

SUMMARY:
Multicenter, randomized, masked, controlled study of the safety and effectiveness of intravitreally administered ONS-5010.

ELIGIBILITY:
Inclusion Criteria:

* Active primary Subfoveal Choroidal Neovascularization lesions secondary to Age-related macular degeneration (AMD) in the study eye
* Best corrected visual acuity of 35-75 letters read (20/32 to 20/200 Snellen equivalent)
* Study eye must:
* Have active leakage on Fluorescein Angiogram involving the fovea
* Have edema involving the fovea
* Be free of scarring, fibrosis, or atrophy involving the central foveal zone

Exclusion Criteria:

* Previous subfoveal focal laser photocoagulation in the study eye
* Laser photocoagulation (juxtafoveal or extrafoveal) in the study eye within 1-month preceding randomization
* Any concurrent intraocular condition in the study eye that may require medical or surgical intervention or contribute to vision loss within 1 year
* Active intraocular inflammation (grade trace or above) in the study eye
* Current vitreous hemorrhage in the study eye
* Polypoidal choroidal vasculopathy (PCV) in the study eye
* History of idiopathic or autoimmune-associated uveitis in either eye
* Infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥30 mmHg despite treatment with anti-glaucoma medication)
* Premenopausal women not using adequate contraception
* Current treatment for active systemic infection
* Known allergy to any component of the study drug or history of allergy to fluorescein , not amenable to treatment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the effectiveness of intravitreal injections of ONS-5010 compared to ranibizumab in preventing vision loss, as measured by the mean change in baseline best correct visual acuity (BCVA) at Week 8 | Baseline, 8 weeks
  BCVA to be assessed as letters read using the Early Treatment Diabetic Retinopathy Study (ETDRS) charts. A positive change represents an improvement in visual acuity.

CONTACTS AND LOCATIONS:
Locations (60):
- United States (60):
  - Clinical Site, Arcadia, California
  - Clinical Site, Bakersfield, California
  - Clinical Site, Beverly Hills, California
  - Clinical Site, Huntington Beach, California
  - Clinical Site, Laguna Hills, California
  - Clinical Site, Long Beach, California
  - Clinical Site, Modesto, California
  - Clinical Site, Oakland, California
  - Clinical Site, Pasadena, California
  - Clinical Site, Poway, California
  - Clinical Site, Sacramento, California
  - Clinical Site, Colorado Springs, Colorado
  - Clinical Site, Lakewood, Colorado
  - Clinical Site, Waterford, Connecticut
  - Clinical Site, Coral Springs, Florida
  - Clinical Site, Fort Lauderdale, Florida
  - Clinical Site, Jacksonville, Florida
  - Clinical Site, Orlando, Florida
  - Clinical Site, Stuart, Florida
  - Clinical Site, Oak Forest, Illinois
  - Clinical Site, Oak Park, Illinois
  - Clinical Site, Carmel, Indiana
  - Clinical Site, Lenexa, Kansas
  - Clinical Site, Lexington, Kentucky
  - Clinical Site, Hagerstown, Maryland
  - Clinical Site, Edina, Minnesota
  - Clinical Site, Saint Louis Park, Minnesota
  - Clinical Site, Jackson, Mississippi
  - Clinical Site, Teaneck, New Jersey
  - Clinical Site, Albuquerque, New Mexico
  - Clinical Site, Liverpool, New York
  - Clinical Site, Oceanside, New York
  - Clinical Site, Rochester, New York
  - Clinical Site, Westbury, New York
  - Clinical Site, Asheville, North Carolina
  - Clinical Site, Hickory, North Carolina
  - Clinical Site, Wake Forest, North Carolina
  - Clinical Site, Winston-Salem, North Carolina
  - Clinical Site, Edmond, Oklahoma
  - Clinical Site, Charleston, South Carolina
  - Clinical Site, Florence, South Carolina
  - Clinical Site, Ladson, South Carolina
  - Clinical Site, West Columbia, South Carolina
  - Clinical Site, Rapid City, South Dakota
  - Clinical Site, Germantown, Tennessee
  - Clinical Site, Abilene, Texas
  - Clinical Site, Arlington, Texas
  - Clinical Site, Austin, Texas
  - Clinical Site, Beaumont, Texas
  - Clinical Site, Bellaire, Texas
  - Clinical Site, Dallas, Texas
  - Clinical Site, Round Rock, Texas
  - Clinical Site, San Antonio, Texas
  - Clinical Site, The Woodlands, Texas
  - Clinical Site, Willow Park, Texas
  - Clinical Site, Salt Lake City, Utah
  - Clinical Site, Fairfax, Virginia
  - Clinical Site, Lynchburg, Virginia
  - Clinical Site, Bellevue, Washington
  - Clinical Site, Silverdale, Washington

IPD SHARING:
Plan to Share IPD: No